CLINICAL TRIAL: NCT05399875
Title: Augmented Reality Ruler to Improve Safety and Clinical Workflow During Placement of Peripherally Inserted Central Catheters
Brief Title: AR Ruler to Improve Safety and Clinical Workflow During PICC Placement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Ali Dhanaliwala, Physician, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 851278
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Insertion of Peripherally Inserted Central Catheter
Keywords: Catheters; Augmented Reality; Radiology, Interventional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Augmented reality virtual ruler (Experimental): Patient's in this arm will have their physician use an augmented reality virtual ruler to measure catheter length during catheter placement.
  Interventions: Other: Augmented reality virtual ruler

INTERVENTIONS:
Other: Augmented reality virtual ruler — Use of augmented reality virtual ruler to measure catheter length

SUMMARY:
The purpose of this study is to assess the utility of an augmented reality virtual ruler during placement of peripherally inserted central catheters.

DETAILED DESCRIPTION:
After being informed about the study, patients who give consent will have their peripheral inserted central catheter placed by a physician wearing mixed reality smart glasses. The mixed reality smart glasses will have an application that allows the physician to measure distances with their hands. This application will be used to measure the appropriate length for which to trim the central catheter.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a non-emergent peripherally inserted central catheter placement in Interventional Radiology
* Over 18 years

Exclusion Criteria:

* Undergoing an emergent peripherally inserted central catheter placement
* Younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with appropriate catheter tip location | End of procedure
  Catheter tip location will be evaluated by the treating physician on x-ray

SECONDARY OUTCOMES:
Radiation dose | End of procedure
  Total radiation dose of the procedure will be captured from the fluoroscopy machine
Procedure time | End of procedure
  Procedure time to complete catheter placement will be captured from the radiology information system.

CONTACTS AND LOCATIONS:
Overall Officials: Ali H Dhanaliwala, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.